CLINICAL TRIAL: NCT01991327
Title: AN OPEN-LABEL, MULTIPLE DOSE STUDY TO ASSESS THE DRUG-DRUG INTERACTIONS OF ANDROXAL WITH CYTOCHROME P450 ISOENZYMES IN HEALTHY MALE SUBJECTS
Brief Title: Assessment of Drug-Drug Interactions of Androxal With Cytochrome P450 Isoenyzmes in Healthy Males
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Repros Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZA-106
Record Dates: First submitted 2013-11-18; First posted 2013-11-25 (Estimated); Last update posted 2014-08-11 (Estimated); Status verified 2014-08

CONDITIONS: Drug-drug Interaction
MeSH Terms: interventions — Enclomiphene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Androxal (Experimental): Androxal 25 mg capsules once a day for 7 days
  Interventions: Drug: Androxal
- Placebo Androxal (Active Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Androxal
  Other Names: enclomiphene citrate
  Arms: Androxal
Drug: Placebo
  Arms: Placebo Androxal

SUMMARY:
The primary objective of this study is to assess the drug-drug interactions of Androxal with cytochrome P450 isoenzymes, CYP1A2, CYP2C8, CYP2C9, CYP2C19, CYP2D6, and CYP3A4 in healthy male subjects administered 25 mg Androxal once daily for 3 days. Secondly, the safety and tolerability of Androxal will be determined in healthy male subjects administered Androxal 25 mg daily for 3 days.

ELIGIBILITY:
Inclusion Criteria:

* Speak, read, and understand English or Spanish and is willing and able to provide written informed consent on an institutional review board (IRB)-approved form prior to the initiation of any study procedures;
* Healthy male, between the ages of 18 and 60 years; body mass index (BMI) 19.0-29.9.
* All laboratory tests either within the normal range or assessed as not clinically significant by the Principal Investigator. Any clinically significant deviations outside of the normal range in the opinion of the Principal Investigator will require sponsor approval. A negative hepatitis B surface antigen, hepatitis C antibody or HIV antibody test result within the previous 3 months may be used instead of obtaining a screening laboratory sample for these laboratory tests;
* Ability to complete the study in accordance with the protocol.

Exclusion Criteria:

* Known hypersensitivity to Clomid;
* A clinically significant laboratory abnormality or other clinical findings indicative of a clinically significant exclusionary disease including hepatic insufficiency, renal insufficiency, unstable coronary artery disease, malignancy other than basal cell carcinoma or squamous cell carcinoma of the skin or stroke;
* A positive hepatitis screen including hepatitis surface B antigen (HBsAg) and hepatitis C antibody;
* A positive test result for HIV;
* Positive results from a urine screen for substances of abuse;
* A recent history of alcoholism (< 2 years) or of moderate alcohol use (greater than an average of 3 drinks per day or a total of 21 drinks per week) or use of alcohol within 24 hours prior to receiving the first dose of study medication;
* Use of any recreational drugs within the past year or a previous history of drug abuse;
* Use of an investigational drug or product, or participation in a drug research study within 30 days prior to receiving study medication;
* A clinically significant electrocardiogram (ECG) abnormality;
* A history of difficulty with phlebotomy;
* Donation of blood (1 pint or more) within 30 days, or plasma within 7 days prior to receiving study medication;
* Use of any prescription drug therapy within 14 days prior to receiving study medication;
* Use of any over-the-counter (OTC) drugs for therapeutic purposes within 48 hours prior to receiving study medication; Use of dietary or herbal supplements 14 days prior to study or megavitamin supplements within 48 hours prior to receiving study medication;
* Consumption of any caffeine containing foods or beverages within 48 hours prior to receiving study medication;
* Consumption of any grapefruit or grapefruit-containing juices, vegetables from the mustard green family, and charbroiled meat within 72 hours prior to receiving study medication;
* Current smoker or user of any tobacco products that has smoked in last 30 or 60 days;
* Any condition which, in the opinion of the Principal Investigator, could interfere with the subject's ability to provide informed consent, comply with study instructions, possibly confound interpretation of study results, or endanger the subject if he took part in the study;
* Classified as a cytochrome P450 isoenzyme 2D6 (CYP2D6) "poor metabolizer" as determined by genotyping at the screening visit
* Use of a monoamine oxidase (MAO) Inhibitor in the previous 28 days prior to dose.
* Concurrent use of cimetidine, levodopa, amantadine, other antipsychotics or antidepressants.
* Type I or Type II diabetes
* Clinical evidence of cirrhosis or biopsy proven cirrhosis of any etiology
* Screening liver function tests (ALT, AST, Bil, Alk. Phos) greater than upper limit of normal
* History of hypertension with BP > 150/95 mmHg seated at screening
* History of chronic pancreatitis or cholelithiasis

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-05; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Drug-Drug Interaction | 3 days
  The primary objective of this study is to assess the drug-drug interactions of Androxal with cytochrome P450 isoenzymes, CYP1A2, CYP2C8, CYP2C9, CYP2C19, CYP2D6, and CYP3A4 in healthy male subjects administered 25 mg Androxal once daily for 3 days.

CONTACTS AND LOCATIONS:
Locations (1):
- Miami, Florida, United States

REFERENCES:
- See also: Sponsor corporate website — http://www.reprosrx.com